CLINICAL TRIAL: NCT02930642
Title: Food Insecurity, Obesity, and Impulsive Food Choice
Acronym: FIOI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IdahoSU001
Record Dates: First submitted 2016-10-05; First posted 2016-10-12 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Feeding Behavior; Obesity; Impulsivity
Keywords: Mindfulness; Obesity; Food insecurity; Delay discounting
MeSH Terms: conditions — Feeding Behavior; Obesity; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindful Eating (Experimental): Participants in this arm will receive a 50 min mindful eating training with four pieces of food. They will practice mindful eating at home with two meals for a one-week duration.
  Interventions: Behavioral: Mindful Eating
- Nutrition Digital Video Disc (DVD) (Active Comparator): Participants will watch a 50 min DVD on nutrition and receive four pieces of food. They will receive prompts twice a week to give one-word answers to questions about food.
  Interventions: Other: Nutrition DVD
- Control (No Intervention): Participants will receive four pieces of food. They will not receive any prompts during the one week.

INTERVENTIONS:
Behavioral: Mindful Eating — Mindful eating is a behavioral strategy in which food is eaten slowly, with deliberate and focused attention on the features of food, the process of eating, and physiological responses to eating. Objectivity is key.
  Other Names: Raisin exercise
  Arms: Mindful Eating
Other: Nutrition DVD — Participants watch a 50 minute video on nutrition to control for verbal aspects of food.
  Arms: Nutrition Digital Video Disc (DVD)

SUMMARY:
The objective of this study is to determine the relations among food insecurity status, obesity, and impulsive food choice patterns and to test the extent to which a mindful eating strategy reduces impulsive choice for food. The central hypothesis is that food-insecure individuals will demonstrate more impulsive food choice patterns and demonstrate a greater likelihood of obesity than individuals who are food secure. Two specific aims are proposed:

Specific aim #1: Determine the relation between food insecurity, obesity, and impulsive food choice patterns in women. The working hypothesis is that food-insecure individuals, especially those that are obese, will exhibit more impulsive food choice patterns than food-secure individuals.

Specific aim #2: Determine the efficacy of an extended mindfulness-based eating strategy on impulsive choice patterns among food insecure women. The working hypothesis is that mindful eating will reduce impulsive food choice patterns relative to baseline and control conditions, and will persist to follow-up. The investigators expect mindful eating to reduce impulsive choice compared to control conditions, despite food security status.

DETAILED DESCRIPTION:
The investigators will recruit women from a variety of community locations, including grocery stores, public schools, churches, local food pantries, and from governmental food assistance programs, such as Women, Infants, and Children and the Supplemental Nutrition Assistance Program. Participants will be recruited heavily from settings where low to moderate food security is prevalent, but not severe food security. Food insecurity status will be determined by completion of the 18-item United State Department of Agriculture (USDA) Food Security Module, and will be scored based on standardized scoring techniques. Participants will provide informed consent, be weighed and measured, and complete several questionnaires that measure diet quality, time since last pay check or food benefits as well as other information, such as age, education, ethnicity, employment status, income, marital status, intelligence, nicotine dependence, and alcohol and drug use. Participants will complete baseline delay and probability discounting tasks for food and money as measures of impulsivity.

Then, food insecure women only will be randomly assigned to one of three arms: mindful eating, a nutrition movie, or a control. Participants in the mindful eating group will be given four foods and receive a 50 min mindful eating workshop. Individuals in the nutrition movie condition also will be given the same four foods, but will view a 50 minute nutrition video. The third group (no treatment control) will receive the four foods, but no treatment. A Time 2 measures of discounting will be administered immediately after the treatments.

Then, for the next week after Session 2, participants in the mindful eating group will be asked to practice mindful eating throughout the week. Research assistants will send text message prompts to participants reminding them to record when they practice mindful eating during meals twice per day for one week. Those in the Nutrition movie will receive the same number of prompts during a one week period as the mindful eating group, but they will give give one-word answers to questions about nutrition. Those in the control group will do nothing during the week.

After one week of mindful eating (or controls), all participants will be asked to return to the laboratory and complete a third set of discounting tasks.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Must be an adult
* Must score 3-5 (with children) or 3-7 (without children) on the USDA Food Security Module
* Must be English speaking

Exclusion Criteria:

* Pregnancy
* Diagnosed with an eating disorder
* HIV
* Hemophilia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Number of impulsive choices as assessed by the Food Choice Questionnaire | Two to three weeks
  Participants will be asked to make a series of hypothetical choices between small, sooner (impulsive) vs. larger, later (self controlled) hypothetical food-related outcomes
Number of impulsive choices as assessed by the Monetary Choice Questionnaire | Two to three weeks
  Participants will be asked to make a series of hypothetical choices between small, sooner (impulsive) vs. larger, later (self controlled) hypothetical monetary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rasmussen, PhD, Principal Investigator — Idaho State University
Locations (1):
- Idaho State University, Pocatello, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lawyer SR, Boomhower SR, Rasmussen EB. Differential associations between obesity and behavioral measures of impulsivity. Appetite. 2015 Dec;95:375-82. doi: 10.1016/j.appet.2015.07.031. Epub 2015 Jul 31. PMID 26235925
- [Background] Rasmussen EB, Lawyer SR, Reilly W. Percent body fat is related to delay and probability discounting for food in humans. Behav Processes. 2010 Jan;83(1):23-30. doi: 10.1016/j.beproc.2009.09.001. Epub 2009 Sep 8. PMID 19744547
- [Background] Hendrickson KL, Rasmussen EB. Effects of mindful eating training on delay and probability discounting for food and money in obese and healthy-weight individuals. Behav Res Ther. 2013 Jul;51(7):399-409. doi: 10.1016/j.brat.2013.04.002. Epub 2013 Apr 27. PMID 23685325
- [Background] Hendrickson KL, Rasmussen EB, Lawyer SR. Measurement and validation of measures for impulsive food choice across obese and healthy-weight individuals. Appetite. 2015 Jul;90:254-63. doi: 10.1016/j.appet.2015.03.015. Epub 2015 Mar 18. PMID 25796210
- [Background] Robaina KA, Martin KS. Food insecurity, poor diet quality, and obesity among food pantry participants in Hartford, CT. J Nutr Educ Behav. 2013 Mar;45(2):159-64. doi: 10.1016/j.jneb.2012.07.001. Epub 2012 Dec 5. PMID 23219294
- [Background] Townsend MS, Peerson J, Love B, Achterberg C, Murphy SP. Food insecurity is positively related to overweight in women. J Nutr. 2001 Jun;131(6):1738-45. doi: 10.1093/jn/131.6.1738. PMID 11385061